CLINICAL TRIAL: NCT06954168
Title: The Effects of Smoking on Sleep Quality, Fatigue and Perceived Stress in University Students: A Comparison Study
Brief Title: The Effects of Smoking on Sleep Quality, Fatigue and Perceived Stress
Status: Not yet recruiting | Type: Observational
Sponsor: Barış SEVEN (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Barış SEVEN, Ph.D, Gazi University
Organization: Gazi University (Other)
Other Study IDs: 7
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-09

CONDITIONS: University Students

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- University students who smoke
- non-smoking university students

SUMMARY:
Tobacco use is a major cause of death resulting from cancer, cardiovascular diseases, and pulmonary disorders. It is also a risk factor for respiratory and other infections, osteoporosis, diabetes, reproductive disorders, adverse surgical outcomes and delayed wound healing, as well as duodenal and gastric ulcers [1]. Studies project that the number of deaths due to smoking will rise to 8.4 million by 2030 [2]. According to the Tobacco Atlas, in Turkey, 83,100 people die each year due to smoking-related causes.

The negative effects of smoking are not limited to chronic diseases; it can also affect the quality of daily life. In a study involving 3,516 participants, it was reported that both male and female smokers experienced significantly greater difficulty falling asleep compared to non-smokers. They also suffered from non-restorative sleep, frequent awakenings during the night, and difficulty falling back asleep [3]. Furthermore, literature has demonstrated a significant relationship between smoking and perceived stress [4]. Perceived stress is defined as "the feelings or thoughts an individual has about how much stress they are under during a particular period" [5]. Although smoking may temporarily alleviate perceived stress, studies suggest it may actually lead to negative emotional states or exacerbate stress in the long run [6, 7]. In addition, it has been found that smokers tend to feel more tired and become fatigued more quickly compared to non-smokers [8, 9].

The majority of smokers begin smoking during adolescence [10]. In their study, Burt et al. reported that 71% of smokers started smoking at or before the age of 18 [11]. The university period is a critical phase in young individuals' lives, and habits formed during this time can have long-term health consequences. Smoking can affect not only health but also academic performance [12]. Factors such as stress [13], sleep quality [14], and fatigue [15], which have previously been studied in smokers, have also been shown to negatively impact academic achievement. Although academic success will not be directly evaluated in our study, considering the target population, the potential secondary effect of smoking on academic performance further underscores the significance of our research.

This study is designed to compare university students who smoke and those who do not in terms of sleep quality, fatigue, and perceived stress levels. Although there are existing studies that examine these parameters individually or in different populations, to our knowledge, no study has simultaneously assessed all of these factors in a university student sample. Most studies in this field focus on the general population; however, university students represent a specific group due to their stressful academic lives, social pressures, and lifestyle changes. The originality of our study lies in its focus on university students and its comprehensive approach to examining multiple variables concurrently. In this context, the planned research will provide more specific and detailed insights into the factors associated with nicotine dependence and their interrelationships.

ELIGIBILITY:
Inclusion Criteria:

* be an actively enrolled undergraduate student

Exclusion Criteria:

* Have a diagnosed sleep disorder such as sleep apnea, insomnia or narcolepsy.
* Have mental health problems such as diagnosed depression, anxiety disorders or bipolar disorder.
* Chronic diseases such as diabetes, hypertension, asthma.
* Conditions that may independently affect sleep, fatigue or stress, such as night shift work and pregnancy.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: University Students
Sampling Method: Probability Sample
Enrollment: 528 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-27 (Estimated)

PRIMARY OUTCOMES:
The Fagerstrom Test for Nicotine Dependence | only once
The Pittsburgh Sleep Quality Index Scoring | only once
The Fatigue Assessment Scale | only once
The Perceived Stress Scale | only once

IPD SHARING:
Plan to Share IPD: No